CLINICAL TRIAL: NCT01580007
Title: Clinical Trial of Oral Phenylbutyrate and Vitamin D Adjunctive Therapy in Pulmonary Tuberculosis in Bangladesh: a Pilot Study
Brief Title: Clinical Trial of Phenylbutyrate and Vitamin D in Tuberculosis (TB)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: International Centre for Diarrhoeal Disease Research, Bangladesh (Other)
Collaborators: Karolinska Institutet (Other); National Institute of Diseases of the Chest and Hospital, Bangladesh (Other); University of Iceland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PR-09068
Record Dates: First submitted 2012-04-17; First posted 2012-04-18 (Estimated); Last update posted 2015-02-13 (Estimated); Status verified 2014-01

CONDITIONS: Pulmonary Tuberculosis
Keywords: tuberculosis; phenylbutyrate; vitamin D; cathelicidin; antimicrobial peptide; in adults
MeSH Terms: conditions — Tuberculosis, Pulmonary; Tuberculosis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Active Sodium Phenylbutyrate and active cholecalciferol (Active Comparator): 500 mg sodium phenylbutyrate (4-phenylbutyric acid, sodium salt) in tablet form twice daily and 5000 IU of cholecalciferol once daily will be given orally for 2 months
  Interventions: Drug: Active Sodium Phenylbutyrate and active cholecalciferol
- Placebo Sodium Phenylbutyrate plus active cholecalciferol (Active Comparator): Drug: Cholecalciferol Placebo: Sodium Phenylbutyrate
  Interventions: Drug: Placebo Sodium Phenylbutyrate plus active cholecalciferol
- Active Sodium Phenylbutyrate and placebo cholecalciferol (Active Comparator): Drug: Sodium Phenylbutyrate Placebo: cholecalciferol
  Interventions: Drug: Active Sodium Phenylbutyrate and placebo cholecalciferol
- Placebo Sodium Phenylbutyrate plus placebo cholecalciferol (Placebo Comparator): Placebo Sodium Phenylbutyrate Placebo cholecalciferol
  Interventions: Drug: Placebo Sodium Phenylbutyrate plus placebo cholecalciferol

INTERVENTIONS:
Drug: Active Sodium Phenylbutyrate and active cholecalciferol — Sodium Phenylbutyrate: 500 mg twice daily orally for 2 months Cholecalciferol: 5000 IU once daily orally for 2 months
  Other Names: triButyrate®; Vigantol oil
  Arms: Active Sodium Phenylbutyrate and active cholecalciferol
Drug: Placebo Sodium Phenylbutyrate plus active cholecalciferol — Placebo Sodium Phenylbutyrate: twice daily orally for 2 months Cholecalciferol: 5000 IU once daily for 2 months
  Other Names: Vigantol oil; Placebo Phenylbutyrate
  Arms: Placebo Sodium Phenylbutyrate plus active cholecalciferol
Drug: Active Sodium Phenylbutyrate and placebo cholecalciferol — Sodium phenylbutyrate: 500 mg twice daily orally for 2 months Placebo cholecalciferol: once daily orally for 2 months
  Other Names: triButyrate®; Placebo vigantol oil
  Arms: Active Sodium Phenylbutyrate and placebo cholecalciferol
Drug: Placebo Sodium Phenylbutyrate plus placebo cholecalciferol — Placebo Sodium Phenylbutyrate: twice daily orally for 2 months Placebo cholecalciferol: once daily orally for 2 months
  Arms: Placebo Sodium Phenylbutyrate plus placebo cholecalciferol

SUMMARY:
Vitamin D exerts its effects via the Vitamin D Receptor (VDR) present in activated macrophages and induces expression and release of the cathelicidin, LL-37, a human antimicrobial peptide involved in killing of MTB. We aimed to investigate whether treatment of newly diagnosed pulmonary TB patients for 2 months with adjunctive PBA and vitamin D (Cholecalciferol) in combination with standard DOTS therapy (i) can improve response to standard short course TB therapy towards a rapid recovery; (ii) can induce expression of LL-37 in macrophages; (iii) can enhance killing capacity of macrophages isolated from TB patients infected in vitro with MTB; and (iv) does not evoke any adverse effects.

DETAILED DESCRIPTION:
This is a double-blind, randomized, placebo controlled clinical trial on clinical efficacy of phenylbutyrate and vitamin D3 therapy daily for 2 months in newly diagnosed sputum smear positive pulmonary TB patients. The clinical trial will take place in the National Institute of the Diseases of the Chest and Hospital (NIDCH) in Dhaka, Bangladesh.

Our specific aims are:

Objective 1: To determine the optimal oral dose of PBA required for induction of antimicrobial peptide in macrophages from healthy adults.

Objective 2

The second aim of this study is to determine whether adjunctive sodium phenylbutyrate and vitamin D treatment (for 2 months) of newly diagnosed pulmonary TB patients:

1. Can improve response to standard short course TB therapy towards a rapid recovery (clinical, radiological, mycobacterial).
2. Can induce expression of LL-37 in macrophages (immunological).
3. Can enhance killing capacity of macrophages from TB patients infected in vitro with MTB (functional measures of treatment outcome).

Study Design: The study will be a randomized, double blind (Subject, Caregiver, Investigator, Outcomes Assessor), placebo control trial for 2 months. It will also be a safety and efficacy phase III study. The study will have a 4x4 factorial design with 4-cell interventions. Enrolled patients will be randomized into the following four treatment arms in a 1:1:1:1 ratio:

Group 1: PBA Group 2: Vitamin D3 (Cholecalciferol) Group 3: PBA plus vitamin D3 Group 4: Placebo

ELIGIBILITY:
Inclusion Criteria:

* Adults, 18-60 years with sputum smear positive pulmonary TB
* New cases only
* Gender, both
* Consent to enroll in the study

Exclusion Criteria:

* Hypercalcaemia (serum calcium > 2.6 mmol/L) identified at baseline
* Taking vitamin D
* Pregnant and lactating
* Any known liver or kidney function abnormality, malignancy

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 288 (Actual)
Dates: Start 2010-12; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Proportion of pulmonary TB patients who are culture negative in sputum in week 4 | week 4
  To determine the proportion of sputum culture positive patients becoming culture negative at 1 and 2 months after adjunctive sodium phenylbutyrate and vitamin D treatment of patients for 2 months.
Difference in improvement in clinical endpoints consisting of cough clearance, percentage chest x-ray clearance, fever remission and weight increase upto 8 weeks. | 8 weeks
  Difference in improvement in clinical endpoints consisting of:
  cough clearance (weekly to week-8 then at week 24) chest x-ray impovement (percentage lung involvement on CXR at week 8) fever remission (weekly to week-8 then at week 24) weight increase (weekly to week-8 then at week 24)

SECONDARY OUTCOMES:
Sputum smear conversion time | weekly up to week 12; then at week 24
Radiological improvement (percent lung involvement on CXR) | week 0, 8, 12 and 24
Cough clearance | weekly up to week 12; then at week 24
Weight gain | weekly up to week 12, then at week 24
Change in plasma PBA concentrations | week 0, 4, 8, 12
Change in plasma 25(OH)D3 concentration | week 0, 4, 8, 12, 24
Clinical failure and default independently and 'death or clinical failure or default' | week 24
Hypercalcaemia (serum calcium > 2.6 mmol/L) | week 0, 2, 4, 8, 12
Gastrointestinal side effects | weekly to week 12 then at week 24
Immunological improvement (LL-37 in macrophages) | week 0, 4, 8, 12
Functional immunological improvement (killing by macrophages) | week 0, 4, 8, 12

CONTACTS AND LOCATIONS:
Locations (1):
- National Institute of Diseases of Chest and Hospital (NIDCH), Dhaka, Bangladesh

REFERENCES:
- [Derived] Rekha RS, Mily A, Sultana T, Haq A, Ahmed S, Mostafa Kamal SM, van Schadewijk A, Hiemstra PS, Gudmundsson GH, Agerberth B, Raqib R. Immune responses in the treatment of drug-sensitive pulmonary tuberculosis with phenylbutyrate and vitamin D3 as host directed therapy. BMC Infect Dis. 2018 Jul 4;18(1):303. doi: 10.1186/s12879-018-3203-9. PMID 29973153
- [Derived] Mily A, Rekha RS, Kamal SM, Arifuzzaman AS, Rahim Z, Khan L, Haq MA, Zaman K, Bergman P, Brighenti S, Gudmundsson GH, Agerberth B, Raqib R. Significant Effects of Oral Phenylbutyrate and Vitamin D3 Adjunctive Therapy in Pulmonary Tuberculosis: A Randomized Controlled Trial. PLoS One. 2015 Sep 22;10(9):e0138340. doi: 10.1371/journal.pone.0138340. eCollection 2015. PMID 26394045
- [Derived] Mily A, Rekha RS, Kamal SM, Akhtar E, Sarker P, Rahim Z, Gudmundsson GH, Agerberth B, Raqib R. Oral intake of phenylbutyrate with or without vitamin D3 upregulates the cathelicidin LL-37 in human macrophages: a dose finding study for treatment of tuberculosis. BMC Pulm Med. 2013 Apr 16;13:23. doi: 10.1186/1471-2466-13-23. PMID 23590701